CLINICAL TRIAL: NCT03674372
Title: Pilot Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in Severe Right and Left Congenital Diaphragmatic Hernia (CDH)
Brief Title: Fetoscopic Endoluminal Tracheal Occlusion
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0461
Record Dates: First submitted 2018-08-24; First posted 2018-09-17 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: tracheal occlusion; FETO; Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Fetuses with Left CDH (O/E LHR < 25%) (Experimental): Fetuses with Left CDH (O/E LHR < 25%) will receive Fetoscopic Endoluminal Tracheal Occlusion (FETO)
  Interventions: Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO)
- Fetuses with L- sided CDH with O/E LHR <30%. (Experimental): Fetuses with Left CDH (O/E LHR < 30%) will receive Fetoscopic Endoluminal Tracheal Occlusion (FETO)
  Interventions: Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO)
- Fetuses with R- sided CDH with O/E LHR < 45% (Experimental): Fetuses with Right CDH (O/E LHR < 45%) will receive Fetoscopic Endoluminal Tracheal Occlusion (FETO)
  Interventions: Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO)

INTERVENTIONS:
Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO) — This study will position and remove an endoluminal tracheal balloon in utero (FETO) to study the feasibility of implementing FETO therapy in the most severe group of fetuses with left CDH (O/E < 25%; O/E LHR < 30 %) and right CDH (O/E LHR < 45%).
  Other Names: BALT GOLDBALLOON: GoldBAL2 Detachable Balloon; BALTACCIBDPE100: Catheter System

SUMMARY:
The purpose of this research study is to see if the FETO surgery and FETO release (surgery to remove the device) works and is safe for babies with severe right or left Congenital Diaphragmatic Hernia (CDH). CDH is a condition in which a hole in the baby's diaphragm allows the abdominal organs to move into the chest and limit lung growth. The goal of the FETO device is to block the airway with a balloon-type device, allowing fluid to build up and help the unborn baby's lungs grow. Bigger lungs may improve the baby's quality of life.

DETAILED DESCRIPTION:
Despite advances in prenatal diagnosis and postnatal therapies, including extracorporeal membrane oxygenation (ECMO), inhaled nitric oxide therapy, and ventilator strategies that minimize ventilator-induced lung injury, morbidity and mortality rates for babies with severe CDH remain high. Data from Children's Hospital of Philadelphia (CHOP) between January 2006 and December 2010 for prenatal and postnatal care for 64 patients with isolated left CDH showed overall survival was 63%. Survival was 33% in patients requiring the use ECMO. Immediate morbidity/mortality is related to the severity of the pulmonary hypoplasia caused by the mass effect of the herniated abdominal contents on the developing lungs. Quantifying the severity of pulmonary hypoplasia has been performed using the observed/expected lung to head circumference ratio (O/E LHR). It is a tool validated in 354 fetuses with unilateral isolated CDH evaluated between 18 and 38 weeks gestation. For O/E LHR < 25%, survival was dismal at 1/9 or 11% (CHOP experience, not published). Published data from an interdisciplinary follow-up program at CHOP shows striking morbidities in neuromuscular tone and neurodevelopmental status.

The rationale for fetal therapy in severe CDH is to improve fetal lung growth and therefore neonatal survival. Prenatal tracheal occlusion obstructs the normal egress of lung fluid during pulmonary development leading to increased lung tissue stretch, increased cell proliferation, and accelerated lung growth. European colleagues have developed foregut endoscopy and techniques to position and remove endoluminal tracheal balloons in utero. Recently, the Belgium group published summary results of FETO showing an improved survival in 175 patients with isolated left CDH from 24% to 49%.

The investigators goal with this pilot study is to study the feasibility of implementing FETO therapy in the most severe group of fetuses with left CDH (O/E< 25%; O/E < 30%) and right CDH (O/E < 45%).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years and older, who are able to consent
* Singleton pregnancy

Fetal

* Normal Karyotype
* Fetal Diagnosis of Isolated Left or Right CDH with liver up
* Gestation at enrollment prior to 29 wks plus 6 days
* SEVERE pulmonary hypoplasia with Ultra Sound L-sided O/E LHR < 25% or R-sided O/E LHR <45%

Exclusion Criteria:

* Pregnant women <18 years of age.
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* Technical limitations precluding fetoscopic surgery
* Rubber latex allergy
* Preterm labor, cervix shortened (<15 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Psychosocial ineligibility, precluding consent
* Inability to remain at FETO site during time period of tracheal occlusion, delivery and postnatal care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Successful placement of Balt Goldbal2 balloon | 7 weeks after placement
  The feasibility of performing the procedure and managing the pregnancy during the period of tracheal occlusion
Successful removal of Balt Goldbal2 balloon | Within 5 weeks prior to delivery
  The feasibility of the removal of the device prior to delivery
Gestational age at delivery | At delivery
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | After Insertion of Balloon to delivery- (from 27 weeks gestational age up to 39 weeks gestational age)
  Incidence of Maternal complications: preterm labor, premature rupture of membranes, oligohydramnios, polyhydramnios, chorioamnionitis)

SECONDARY OUTCOMES:
Survival at Discharge or at 6 months if still hospitalized | Discharge up to 180 days post delivery
Lung Volume Measurement | 7 weeks after placement of balloon
Lung Head Ratio Measurement | 7 weeks after placement of balloon

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Claus F, Sandaite I, DeKoninck P, Moreno O, Cruz Martinez R, Van Mieghem T, Gucciardo L, Richter J, Michielsen K, Decraene J, Devlieger R, Gratacos E, Deprest JA. Prenatal anatomical imaging in fetuses with congenital diaphragmatic hernia. Fetal Diagn Ther. 2011;29(1):88-100. doi: 10.1159/000320605. Epub 2010 Nov 9. PMID 21063073
- [Background] Danzer E, Gerdes M, Bernbaum J, D'Agostino J, Bebbington MW, Siegle J, Hoffman C, Rintoul NE, Flake AW, Adzick NS, Hedrick HL. Neurodevelopmental outcome of infants with congenital diaphragmatic hernia prospectively enrolled in an interdisciplinary follow-up program. J Pediatr Surg. 2010 Sep;45(9):1759-66. doi: 10.1016/j.jpedsurg.2010.03.011. PMID 20850617
- [Background] Deprest JA, Hyett JA, Flake AW, Nicolaides K, Gratacos E. Current controversies in prenatal diagnosis 4: Should fetal surgery be done in all cases of severe diaphragmatic hernia? Prenat Diagn. 2009 Jan;29(1):15-9. doi: 10.1002/pd.2108. No abstract available. PMID 19125386
- [Background] Luks FI, Deprest JA, Vandenberghe K, Laermans I, De Simpelaere L, Brosens IA, Lerut T. Fetoscopy-guided fetal endoscopy in a sheep model. J Am Coll Surg. 1994 Jun;178(6):609-12. PMID 8193755
- [Background] Deprest J, Nicolaides K, Done' E, Lewi P, Barki G, Largen E, DeKoninck P, Sandaite I, Ville Y, Benachi A, Jani J, Amat-Roldan I, Gratacos E. Technical aspects of fetal endoscopic tracheal occlusion for congenital diaphragmatic hernia. J Pediatr Surg. 2011 Jan;46(1):22-32. doi: 10.1016/j.jpedsurg.2010.10.008. PMID 21238635
- [Background] Deprest J, Gratacos E, Nicolaides KH; FETO Task Group. Fetoscopic tracheal occlusion (FETO) for severe congenital diaphragmatic hernia: evolution of a technique and preliminary results. Ultrasound Obstet Gynecol. 2004 Aug;24(2):121-6. doi: 10.1002/uog.1711. PMID 15287047
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Harrison MR, Adzick NS, Flake AW, VanderWall KJ, Bealer JF, Howell LJ, Farrell JA, Filly RA, Rosen MA, Sola A, Goldberg JD. Correction of congenital diaphragmatic hernia in utero VIII: Response of the hypoplastic lung to tracheal occlusion. J Pediatr Surg. 1996 Oct;31(10):1339-48. doi: 10.1016/s0022-3468(96)90824-6. PMID 8906657
- [Background] Flake AW, Crombleholme TM, Johnson MP, Howell LJ, Adzick NS. Treatment of severe congenital diaphragmatic hernia by fetal tracheal occlusion: clinical experience with fifteen cases. Am J Obstet Gynecol. 2000 Nov;183(5):1059-66. doi: 10.1067/mob.2000.108871. PMID 11084541
- [Background] Harrison MR, Mychaliska GB, Albanese CT, Jennings RW, Farrell JA, Hawgood S, Sandberg P, Levine AH, Lobo E, Filly RA. Correction of congenital diaphragmatic hernia in utero IX: fetuses with poor prognosis (liver herniation and low lung-to-head ratio) can be saved by fetoscopic temporary tracheal occlusion. J Pediatr Surg. 1998 Jul;33(7):1017-22; discussion 1022-3. doi: 10.1016/s0022-3468(98)90524-3. PMID 9694087
- [Background] Harrison MR, Sydorak RM, Farrell JA, Kitterman JA, Filly RA, Albanese CT. Fetoscopic temporary tracheal occlusion for congenital diaphragmatic hernia: prelude to a randomized, controlled trial. J Pediatr Surg. 2003 Jul;38(7):1012-20. doi: 10.1016/s0022-3468(03)00182-9. PMID 12861529
- [Background] Harrison MR, Keller RL, Hawgood SB, Kitterman JA, Sandberg PL, Farmer DL, Lee H, Filly RA, Farrell JA, Albanese CT. A randomized trial of fetal endoscopic tracheal occlusion for severe fetal congenital diaphragmatic hernia. N Engl J Med. 2003 Nov 13;349(20):1916-24. doi: 10.1056/NEJMoa035005. PMID 14614166
- [Background] Benachi A, Chailley-Heu B, Delezoide AL, Dommergues M, Brunelle F, Dumez Y, Bourbon JR. Lung growth and maturation after tracheal occlusion in diaphragmatic hernia. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):921-7. doi: 10.1164/ajrccm.157.3.9611023. PMID 9517613
- [Background] De Paepe ME, Johnson BD, Papadakis K, Sueishi K, Luks FI. Temporal pattern of accelerated lung growth after tracheal occlusion in the fetal rabbit. Am J Pathol. 1998 Jan;152(1):179-90. PMID 9422535
- [Background] Bratu I, Flageole H, Laberge JM, Chen MF, Piedboeuf B. Pulmonary structural maturation and pulmonary artery remodeling after reversible fetal ovine tracheal occlusion in diaphragmatic hernia. J Pediatr Surg. 2001 May;36(5):739-44. doi: 10.1053/jpsu.2001.22950. PMID 11329579
- [Background] Davey MG, Hedrick HL, Bouchard S, Mendoza JM, Schwarz U, Adzick NS, Flake AW. Temporary tracheal occlusion in fetal sheep with lung hypoplasia does not improve postnatal lung function. J Appl Physiol (1985). 2003 Mar;94(3):1054-62. doi: 10.1152/japplphysiol.00733.2002. PMID 12571135
- [Background] Bratu I, Flageole H, Laberge JM, Possmayer F, Harbottle R, Kay S, Khalife S, Piedboeuf B. Surfactant levels after reversible tracheal occlusion and prenatal steroids in experimental diaphragmatic hernia. J Pediatr Surg. 2001 Jan;36(1):122-7. doi: 10.1053/jpsu.2001.20027. PMID 11150450
- [Background] Flageole H, Evrard VA, Piedboeuf B, Laberge JM, Lerut TE, Deprest JA. The plug-unplug sequence: an important step to achieve type II pneumocyte maturation in the fetal lamb model. J Pediatr Surg. 1998 Feb;33(2):299-303. doi: 10.1016/s0022-3468(98)90451-1. PMID 9498406
- [Background] Done E, Gucciardo L, Van Mieghem T, Jani J, Cannie M, Van Schoubroeck D, Devlieger R, Catte LD, Klaritsch P, Mayer S, Beck V, Debeer A, Gratacos E, Nicolaides K, Deprest J. Prenatal diagnosis, prediction of outcome and in utero therapy of isolated congenital diaphragmatic hernia. Prenat Diagn. 2008 Jul;28(7):581-91. doi: 10.1002/pd.2033. PMID 18634116